CLINICAL TRIAL: NCT02197169
Title: A Phase 1b, Randomized, Multi-center, Open-label Study of a Conditionally Replicative Adenovirus (DNX-2401) and Interferon Gamma (IFN-γ) for Recurrent Glioblastoma or Gliosarcoma (TARGET-I)
Brief Title: DNX-2401 With Interferon Gamma (IFN-γ) for Recurrent Glioblastoma or Gliosarcoma Brain Tumors
Acronym: TARGET-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DNAtrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2401BT-IFN-001
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Glioblastoma or Gliosarcoma
Keywords: Brain; Brain Cancer; Brain Neoplasms; Central Nervous System Diseases; Central Nervous System Neoplasms; CNS; Conditionally Replication-Competent Adenovirus; DNX-2401; Delta-24-RGD; Glioma; Glioblastoma; Gliosarcoma; Interferon gamma; Malignant brain tumor; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Nervous System Diseases; Alcyone Lifesciences; AMC™; Cannula; Alcyone MEMS Cannula (AMC™) System
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Central Nervous System Diseases; Central Nervous System Neoplasms; Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Nervous System Diseases | interventions — Oncolytic Virotherapy; Interferon-gamma; interferon gamma-1b; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DNX-2401 alone (Experimental): Single intratumoral injection of DNX-2401
  Interventions: Drug: Single intratumoral injection of DNX-2401
- DNX-2401 + Interferon gamma (IFN-γ) (Experimental): Interferon gamma (IFN-γ) beginning at Day 14
  Interventions: Drug: Single intratumoral injection of DNX-2401; Drug: Interferon-gamma

INTERVENTIONS:
Drug: Single intratumoral injection of DNX-2401 — In the randomized group, following brain tumor biopsy and histological confirmation of recurrent glioblastoma/gliosarcoma, a single injection of DNX-2401 was administered directly into the brain tumor with or without subsequent interferon gamma (IFN-γ)
  No additional subjects will be randomized. A single intratumoral dose of DNX-2401 will be delivered by cannula.
  Other Names: Oncolytic virus; Genetically-modified adenovirus
Drug: Interferon-gamma — In the randomized group, a single injection of DNX-2401 was followed by interferon gamma (IFN-γ). No additional subjects will be randomized or receive IFN-γ following DNX-2401
  Other Names: Actimmune; immunotherapy; gamma interferon
  Arms: DNX-2401 + Interferon gamma (IFN-γ)

SUMMARY:
Glioblastoma (GBM) and gliosarcoma (GS) are the most common and aggressive forms of malignant primary brain tumor in adults and can be resistant to conventional therapies. The purpose of this Phase Ib study is to evaluate how well a recurrent glioblastoma or gliosarcoma tumor responds to one injection of DNX-2401, a genetically modified, conditionally replicative and oncolytic human-derived adenovirus. DNX-2401 is delivered directly into the tumor where it may establish an active infection by replicating in and killing tumor cells.

DETAILED DESCRIPTION:
Enrollment has been completed for the randomized portion of the study with ongoing evaluation of tumor response and safety. No additional subjects will be randomized or receive interferon gamma (IFN-γ).

The non-randomized portion of the study is open for screening and enrollment. Eligible subjects will receive a single intratumoral injection of DNX-2401 into a recurrent glioblastoma or gliosarcoma brain tumor using the Alcyone MEMS Cannula (AMC™) System (cannula). Tumor response and safety will be evaluated.

After receiving DNX-2401, subjects will return to the clinic for study visits at regular intervals for safety monitoring, MRI scans and other assessments for up to 18 months. Thereafter, they will be followed closely for safety and survival.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma or gliosarcoma in first or second recurrence only
* Documented tumor recurrence or progression after failing prior surgical resection, chemotherapy, or radiation
* Tumor size greater than or equal to 1.0 cm in two perpendicular diameters
* Not undergoing surgical resection or for whom gross total resection is not possible
* Karnofsky Performance Status greater than or equal to 70%

Exclusion Criteria:

* Multiple intracranial malignant glioma lesions
* Tumor location or involvement that would result in risk of ventricular penetration during tumor injection
* Tumor involving both hemispheres or that which involves the subependyma or suspected cerebrospinal fluid dissemination
* Tumor involving brain stem
* Documented extracranial metastasis
* Inability to undergo MRI
* Pregnant or nursing females
* Any medical condition that precludes the surgery necessary to administer DNX-2401 into the tumor using the cannula
* Immunocompromised subjects or those with autoimmune conditions, active hepatitis or positive for human immunodeficiency virus (HIV)
* Li-Fraumeni Syndrome

Other protocol-defined inclusion/exclusion criteria may apply as outlined in the relevant protocol version

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) determined by MRI scan review | 1.5 years
  Interval tumor size change will be measured

SECONDARY OUTCOMES:
Incidence and severity of adverse events, including changes in laboratory test results and neurological examination findings | 1.5 years
  Events are classified using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Number of subjects with immunological and biological effects after DNX-2401 with Interferon gamma | 1.5 years
  Laboratory test results and other assessments will be utilized to determine effects
Changes in steroid use (dose and frequency) and clinical and KPS status overall and per study arm assignment | 1.5 years
Overall survival (OS), progression-free survival (PFS), and clinical benefit rate (CBR). | 1.5 years
Changes in responses to quality of life questionnaires | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nam Tran, MD, PhD, Principal Investigator — Moffitt Cancer Center; Karen Fink, MD, PhD, Principal Investigator — Baylor University: Charles A. Sammons Cancer Center; Vinay Puduvalli, MBBS, Principal Investigator — Ohio State University: James Cancer Center; Frederick Lang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - The Ohio State University, Columbus, Ohio
  - Baylor University: Charles A. Sammons Cancer Center, Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas